CLINICAL TRIAL: NCT02674191
Title: Evaluation of Posterior Segment Intrusion Using Miniplates in Skeletal ClassII Hyperdivergent Adolescence: A Randomized Control Trial
Brief Title: Posterior Segment Intrusion Using Miniplates
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Manal El Namrawy (Other)
Responsible Party: Sponsor-Investigator, Manal El Namrawy, assistant lecturer, Cairo University
Organization: Cairo University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Jan 2016. Version 1
Record Dates: First submitted 2016-01-29; First posted 2016-02-04 (Estimated); Last update posted 2018-02-23 (Actual); Status verified 2018-02

CONDITIONS: Orthodontic Anchorage Procedures
Keywords: miniplates ,molar intrusion, hyperdivergent
MeSH Terms: interventions — WW Domain-Containing Oxidoreductase; Clindamycin; Diclofenac; Anti-Inflammatory Agents, Non-Steroidal

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Experimental): Device: mini-plates supported molar intrusion (Stryker, Leibinger, GmbH& Co., Freiburg, Germany) for molar intrusion using miniplates to treat hyperdivergent adolescence Procedure/Surgery: Application of ULTRACARE benzocaine 20%, topical anesthesia (Ultradent Products, Inc) Procedure/Surgery: Administration of , Mepivacaine-l local anesthesia Procedure/Surgery: BETADINE povidone-iodine 10% a local disinfectant Drug: (150g Clindamycin/tds) for 1 week Postoperative antibiotic Drug: (Cataflam 25mg), are prescribed post-operatively an analgesic
  Interventions: Device: mini-plates supported molar intrusion; Procedure: Application of ULTRACARE benzocaine 20%,; Procedure: Administration of , Mepivacaine-l; Procedure: BETADINE povidone-iodine 10%; Drug: (150g Clindamycin/tds) for 1 week; Drug: (Cataflam 25mg), are prescribed post-operatively
- Group 2 (No Intervention): hyperdivergent adolescence with no intervention

INTERVENTIONS:
Device: mini-plates supported molar intrusion — (Stryker, Leibinger, GmbH& Co., Freiburg, Germany) for molar intrusion using miniplates to treat hyperdivergent adolescence
  Arms: Group 1
Procedure: Application of ULTRACARE benzocaine 20%, — topical anesthesia (Ultradent Products, Inc)
  Arms: Group 1
Procedure: Administration of , Mepivacaine-l — local anesthesia
  Arms: Group 1
Procedure: BETADINE povidone-iodine 10% — a local disinfectant
  Arms: Group 1
Drug: (150g Clindamycin/tds) for 1 week — Postoperative antibiotic
  Other Names: Dalacin
  Arms: Group 1
Drug: (Cataflam 25mg), are prescribed post-operatively — an analgesic
  Other Names: NSAIDs
  Arms: Group 1

SUMMARY:
Treating hyperdivergent malocclusion accompanied by open bite could be challenging and may be done by several methods as high pull headgear and posterior bite planes or surgically by maxillary impaction in adults. Nowadays it's the skeletal anchorage system (SAS) era as mini-screws and mini-plates ,hence we are aiming for absolute anchorage, and could minimize patient cooperation and the need for surgical treatment.

DETAILED DESCRIPTION:
Interventions:

A. Treatment group:

Medical History Questionnaire: will be filled by the patient to exclude the presence of any systemic condition.

Clinical Examination:

Oral structures will be examined by (M. N.) including Teeth for caries, fracture or missing teeth and gingival tissues for gingivitis, periodontitis, attachment loss, gingival recession, oral lesions and the nature of the gingival biotype.

The thorough intraoral examination is needed to evaluate the need for referral for consultation or intervention before the initiation of treatment.

Diagnosis: (M. B.) will check the patient to fulfill the previously mentioned inclusion criteria.

Full set of records will be taken for every patient as part of the routine procedure for treatment of patients in the outpatient clinic of the Orthodontic Department, Cairo University.

Clinical Procedures:

The clinical procedures are to be performed according to the protocol applied by Sherwood et al

1. Patients will be referred for the uptake of a Cone Beam Computed Tomography (CBCT), which is considered as (T1). CBCT scanning will be performed with patients in maximum dental intercuspation with the next generation i-CAT CBCT unit according to the manufacture instructions.

   During scanning, the patient position will be standardized as follows; the Frankfort horizontal plane is parallel to the floor and mid sagittal plane is perpendicular to the Frankfort horizontal plane.
2. Banding of the upper first molars will be done followed by taking an upper impression with the molar bands in place.

   A Transpalatal arch (TPA) will be fabricated from 0.9 mm wire and cemented in the upper arch. Bonding of the posterior segment with 3M brackets with MBT prescription 0.022" slot bracket system will be performed. Passive arch of 0.019×0.025" stainless steel arch wire will be placed in the posterior segment bilaterally
3. Surgical procedures will be performed by (H. A.) and will include the following:

   Application of topical anesthesia, ULTRACARE benzocaine 20%, at the local anesthesia injection sites. Administration of local anesthesia, Mepivacaine-l. The injection will be infiltrated into the area where the miniplate will be fixed bilaterally. Proper disinfection will be performed with a local disinfectant, BETADINE povidone-iodine 10%, at the area. Surgery begins with a 1- to 2-cm vestibular incision and a full-thickness mucoperiosteal flap reflected to expose the cortical bone of the maxillary strut by blade no. 15 mounted on Bard Parker handle no.3. Two long Y or I shaped mini plates will be placed bilaterally at the zygomatic buttress area under local anesthesia. The mini plates will be adapted to fit the contour the underlying bone and adjusted to have their terminal part at the upper first molar area. Drilling is done using compatible sized drills mounted on low-speed air motor to create three holes at the sites of the mini screws that will be inserted for fixation of the mini plates.

   The mini plates will be fixed by three mini screws (diameter of 2 mm and 10 mm length) made of titanium. In case of loose mini screws upon tapping, emergency screws will be used instead of the loose ones (wider diameter so will enhance the interlocking with bone).

   After placement of the right and left miniplates, the flap was closed using black silk (3/0) continuous sutures leaving the extensions of the plates perforating the attached gingiva near the mucogingival junction.

   Postoperative instructions will be given to the patients, ice packs, a soft diet is advised. Postoperative antibiotic (150g Clindamycin/tds) for 1 week, as well as an analgesic (Cataflam 25mg), are prescribed post-operatively.

   Strict Oral hygiene instructions will be given to the patients and they will be recalled 1 week after the procedure to ensure adequate soft tissue healing. Sutures are removed one week after the surgery.
4. Closed coil spring insertion:

   Loading of the mini plates was done three weeks after surgery to allow giving sufficient time for soft tissue healing. An intrusion force of (200-300) gm. produced by stretched closed coil spring will be applied and measured by a force gauge .
5. Follow up period:

   The patient will be asked to attend follow-up visits every 4 weeks to check the following: by (M. B., F.H., and M. N.) The stability of the mini plates The integrity of the appliances The activity of the appliance The amount of correction achieved Any inflammation related to the appliance or the mini plates
6. Appliance activation: The appliance will be activated every 4 weeks by (M. N.)
7. The patients of both groups were asked to mark their degree of pain on a (VAS) visual analogue scale regarding their experience with the treatment phase.
8. Termination and intervention: (The end point)

   * Reaching adequate overbite and inter-labial gap or 6 month from the start of intervention
   * Patient request
   * Poor oral hygiene
   * Abnormal side effects or severe inflammation
9. Post-intrusion:

   A second records image will be ordered with the same criteria and parameters as previously mentioned. It is recorded as T2.
10. Patients are going to continue treatment for existing malocclusion and for final detailing of occlusion

Criteria for modifying the allocated intervention:

In case of prolonged swelling and/or pain related to the mini plates, the patient might wait for more than three weeks before coil spring insertion.

In case of loose or broken mini plates, surgical intervention may be required for replacement of the mini plates and the treatment can be resumed after total resolution of the inflammation.

Adherence:

The patients will be asked to attend regular follow-up visits and their adherence to the appointments will be regularly monitored. Reminder calls or messages will be utilized to improve adherence. The patient adherence to intervention instructions will be monitored.

All the participants will be included in an intention to treat analysis, regardless of adherence.

B. Control group:

The subjects should be fulfilling the previously mentioned inclusion criteria and should sign the informed consent of agreement to be recruited in the study.

According to the randomization sheet (done by E.M.), the patients allocated to the control group will be immediately referred for the uptake of a CBCT, which will be considered (T1) without any treatment procedures.

A "no treatment" phase of 6 months will be carried out through which the patients will be followed up to monitor any factor that might have occurred to exclude the patient from the study.

Another CBCT image will be taken after 6 months (T2), T2 images are to be considered the initial diagnostic images for the patient. The patients will then assessed and treatment will be provided for each patient as required.

Adherence:

The patients will be asked to attend regular follow-up visits in which full intra oral and extra oral examination will be performed (E.M.and M.N). Referral of the patient for restorative and/or periodontal therapy may be done with the needs of each case. The patients' adherence to the appointments will be regularly monitored. Reminder calls or messages will be utilized to improve adherence.

. Patients in the control group are going to start treatment for their existing malocclusion by (M. N)

Participant timeline:

The patients will be requested to visit the institutional clinic doing the required adjustments during the preparatory phase

The patients will then be scheduled to attend on the day of surgery, 1 week, 2 and 3 weeks after the surgery. They will also be requested for immediate show up in cases of emergency.

During posterior segment intrusion, the patients will be scheduled to attend every 3-4 weeks for appliance activation and monitoring the treatment progress.

The control group patients will be requested to visit the clinic every 4 weeks for follow up and improvement of the patients' adherence.

ELIGIBILITY:
Inclusion Criteria:

* Mild to moderate skeletal Class II
* Super eruption of maxillary posterior segment
* Erupted full set of maxillary permanent teeth except 3rd molar
* Increased lower facial height

Exclusion Criteria:

* Previous orthodontic treatment

  * Any hormonal disorders or syndromes
  * Systemic Disease
  * Facial Asymmetry
  * Para-functional habits

Ages: 14 Years to 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 24 (Actual)
Dates: Start 2016-05 (Actual); Primary Completion 2018-06 (Estimated); Study Completion 2018-07 (Estimated)

PRIMARY OUTCOMES:
Lower facial height: the distance between soft tissue subnasale and gnathion (Sn.Gn) the difference will be measured in mm. before and after posterior segment intrusion | 6 months
  This measurement relates principally to the vertical dimensions of the upper dento-alveolar process and the mandible.

CONTACTS AND LOCATIONS:
Overall Officials: Manal M El Namrawy, MSc., Principal Investigator — assistant lecturer , Beni suef university

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Kuroda S, Sakai Y, Tamamura N, Deguchi T, Takano-Yamamoto T. Treatment of severe anterior open bite with skeletal anchorage in adults: comparison with orthognathic surgery outcomes. Am J Orthod Dentofacial Orthop. 2007 Nov;132(5):599-605. doi: 10.1016/j.ajodo.2005.11.046. PMID 18005833
- [Background] Ng J, Major PW, Flores-Mir C. True molar intrusion attained during orthodontic treatment: a systematic review. Am J Orthod Dentofacial Orthop. 2006 Dec;130(6):709-14. doi: 10.1016/j.ajodo.2005.05.049. PMID 17169732
- [Result] Sherwood KH, Burch JG, Thompson WJ. Closing anterior open bites by intruding molars with titanium miniplate anchorage. Am J Orthod Dentofacial Orthop. 2002 Dec;122(6):593-600. doi: 10.1067/mod.2002.128641. PMID 12490869
- [Result] Greenlee GM, Huang GJ, Chen SS, Chen J, Koepsell T, Hujoel P. Stability of treatment for anterior open-bite malocclusion: a meta-analysis. Am J Orthod Dentofacial Orthop. 2011 Feb;139(2):154-69. doi: 10.1016/j.ajodo.2010.10.019. PMID 21300243
- [Result] Xun C, Zeng X, Wang X. Microscrew anchorage in skeletal anterior open-bite treatment. Angle Orthod. 2007 Jan;77(1):47-56. doi: 10.2319/010906-14R.1. PMID 17029531